CLINICAL TRIAL: NCT03079713
Title: Comparison of Handheld Vibrator to Topical Eye Drops as Anesthesia for Intravitreal Injections
Brief Title: Handheld Vibrator Versus Topical Eye Drops as Anesthesia for Intravitreal Injections
Acronym: Eyebrator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Dr Mitchell Fineman MD, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-600E
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Pain Control During Intravitreal Injections
Keywords: pain; anesthesia; vibrator; intravitreal; injection
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vibratory Anesthesia (Experimental): Following administration of topical anesthetic and betadine, wearable vibrator will be triggered prior to and during the intravitreal injection
  Interventions: Device: Handheld vibrator triggered during intravitreal injection for wet ARMD
- Standard Injection. (Sham Comparator): Following administration of topical anesthetic and betadine, wearable vibrator will be placed against the lower lid but NOT triggered prior to and during the intravitreal injection
  Interventions: Device: Handheld vibrator not triggered during intravitreal injection for wet ARMD
- Vibratory Anesthesia with Corneal/Conjunctival Sensation Test (Experimental): Healthy patients not requiring intravitreal injection will be subjected to corneal and conjunctival aesthesiometry with and without the vibrator triggered while in contact with the lower eyelid of a single eye.
  Interventions: Device: Normal eye esthesiometry with and without vibration

INTERVENTIONS:
Device: Handheld vibrator triggered during intravitreal injection for wet ARMD — A vibratory device cleaned with alcohol swabs between each use will be attached to the injectors' finger, placed on the lower eyelid of the treatment eye, and triggered during intravitreal injection
  Arms: Vibratory Anesthesia
Device: Normal eye esthesiometry with and without vibration — Healthy patients will undergo corneal and conjunctival esthesiometry with and without triggering of the wearable vibrator placed upon the lower lid of a single eye.
  Arms: Vibratory Anesthesia with Corneal/Conjunctival Sensation Test
Device: Handheld vibrator not triggered during intravitreal injection for wet ARMD — Control group undergoing standard intravitreal injection without triggering of the vibrator.
  Arms: Standard Injection.

SUMMARY:
Intravitreal injections are an efficient method of delivering therapeutic levels of medications to the posterior segment of the eye. Prior to receiving an injection, there are various methods to provide ocular anesthesia. Vibration may have an anti-nociceptive effect by directly decreasing the sensitivity of peripheral nociceptors or by reducing signal transmission from peripheral nociceptors to the brain with activation of vibratory sensation pathways. The purpose of this study is to evaluate the use of a handheld fingertip vibrator compared to topical eye drops for pain control while performing intravitreal eye injections. A secondary objective of the study is to measure corneal and conjunctiva sensitivity with and without activation of the vibrator to the lower lid using a Luneau Cochet-Bonnet aesthesiometer.

DETAILED DESCRIPTION:
A total of 80 patients will be recruited for part 1 of the study. Participants will be randomized in a 1:1 ratio to a standard anesthetic group or standard anesthetic with vibration groups. All intravitreal drugs will be delivered via 30 gauge needles through the pars plana in the inferotemporal quadrant 3.5 to 4 mm posterior to the limbus. Once recruited, a single eye requiring injection for each enrolled patient will be randomized into 1 of 2 groups: aesthesiometer measurement alone with sham vibration (vibrator will not be triggered) (Group 1) or handheld vibrator application and triggering followed by aesthesiometer measurement (Group 2). The vibrator will be applied to the lower eyelid while retracting it during standard intravitreal injection prepped with topical anesthetic (Proparacaine 1%) and Betadine. The main outcome measure of will be patient comfort, as measured by the patient using a standardized Wong-Baker FACES Pain Rating Scale.

An additional 30 eyes of 30 healthy patients not requiring intravitreal injection will be recruited to determine the effect of vibrator application and triggering to the lower lid on corneal and conjunctival (inferotemporal quadrant) sensation as measured using an aesthesiometer. No topical anesthetic will be applied prior to esthesiometry measurements are taken with and without vibration triggering.

All patient identifying information will be removed and patients will be identified with a random number. Data will be checked regularly by a data monitoring committee. Patient records will be reviewed and the following data will be collected: demographic data (age, gender, injected eye, reason for injection), best-corrected visual acuity, intraocular pressure, and complications/adverse events associated with intravitreal injections. Statistical analyses will include univariate comparisons between treatment groups using the Student t-test for continuous variables and χ2 test or Fisher's exact test for categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of neovascular age related macular degeneration requiring anti-VEGF intravitreal injection in the routine course of their care

Exclusion Criteria:

* History of endophthalmitis, prior ocular surgery except cataract surgery, globe rupture, retinal detachment, neurotrophic keratopathy, a history of corneal epithelial basement membrane dystrophy, recent corneal abrasion or trauma, history of infectious keratitis, lower eyelid pathology, those with a previously documented hypersensitivity to ophthalmic 5% povidone-iodine solution (Betadine; Alcon Labs, Fort Worth, TX) or inability to grade pain using the pain scale, pregnant patients, institutionalized patients (nursing home residents, prisoners), those with a history of diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-01-24 (Actual); Study Completion 2019-03-20 (Actual)

PRIMARY OUTCOMES:
Pain assessment | Immediately after intravitreal injection
  Pain is assessed by Wong-Baker FACES Pain Rating Scale (score ranging from 0 to 10) immediately after the intravitreal injection

SECONDARY OUTCOMES:
Corneal and conjunctival sensitivity | immediately after application of a handheld vibrator
  Corneal and conjunctival sensitivity, as measured using an aesthesiometer

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Fineman, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- MidAtlantic Retina-Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman SM, Margo CE. Topical gel vs subconjunctival lidocaine for intravitreous injection: a randomized clinical trial. Am J Ophthalmol. 2006 Nov;142(5):887-8. doi: 10.1016/j.ajo.2006.06.033. PMID 17056383
- [Background] Kaderli B, Avci R. Comparison of topical and subconjunctival anesthesia in intravitreal injection administrations. Eur J Ophthalmol. 2006 Sep-Oct;16(5):718-21. doi: 10.1177/112067210601600509. PMID 17061223
- [Background] Cintra LP, Lucena LR, Da Silva JA, Costa RA, Scott IU, Jorge R. Comparative study of analgesic effectiveness using three different anesthetic techniques for intravitreal injection of bevacizumab. Ophthalmic Surg Lasers Imaging. 2009 Jan-Feb;40(1):13-8. doi: 10.3928/15428877-20090101-05. PMID 19205490
- [Background] Karabas VL, Ozkan B, Kocer CA, Altintas O, Pirhan D, Yuksel N. Comparison of two anesthetic methods for intravitreal ozurdex injection. J Ophthalmol. 2015;2015:861535. doi: 10.1155/2015/861535. Epub 2015 Apr 9. PMID 25949822
- [Background] Ornek N, Apan A, Ornek K, Gunay F. Anesthetic effectiveness of topical levobupivacaine 0.75% versus topical proparacaine 0.5% for intravitreal injections. Saudi J Anaesth. 2014 Apr;8(2):198-201. doi: 10.4103/1658-354X.130713. PMID 24843332
- [Background] Lundeberg TC. Vibratory stimulation for the alleviation of chronic pain. Acta Physiol Scand Suppl. 1983;523:1-51. PMID 6609524
- [Background] Smith KC, Comite SL, Balasubramanian S, Carver A, Liu JF. Vibration anesthesia: a noninvasive method of reducing discomfort prior to dermatologic procedures. Dermatol Online J. 2004 Oct 15;10(2):1. PMID 15530291
- [Background] Aminabadi NA, Farahani RM, Balayi Gajan E. The efficacy of distraction and counterstimulation in the reduction of pain reaction to intraoral injection by pediatric patients. J Contemp Dent Pract. 2008 Sep 1;9(6):33-40. PMID 18784857
- [Background] Bagherian A, Sheikhfathollahi M. Children's behavioral pain reactions during local anesthetic injection using cotton-roll vibration method compared with routine topical anesthesia: A randomized controlled trial. Dent Res J (Isfahan). 2016 May-Jun;13(3):272-7. doi: 10.4103/1735-3327.182189. PMID 27274349
- [Background] Nanitsos E, Vartuli R, Forte A, Dennison PJ, Peck CC. The effect of vibration on pain during local anaesthesia injections. Aust Dent J. 2009 Jun;54(2):94-100. doi: 10.1111/j.1834-7819.2009.01100.x. PMID 19473149